CLINICAL TRIAL: NCT00100100
Title: Modafinil for the Treatment of Cocaine Dependence
Brief Title: Modafinil for the Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Liza Gorgon, National Institute on Drug Abuse
Purpose: Diagnostic
Other Study IDs: NIDA-MDS-0004-1
Record Dates: First submitted 2004-12-22; First posted 2004-12-23 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-07

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of modafinil in reducing cocaine use in subjects with cocaine dependence.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, parallel group design study to evaluate the efficacy and safety of modafinil in reducing cocaine use in subjects with cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have DSM-IV diagnosis of cocaine dependence as determined by SCID.
* Must be seeking treatment for cocaine dependence.
* Must be able to understand and provide written informed consent.

Exclusion Criteria:

* Please contact the study site for more information.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 2004-10; Study Completion 2006-12

PRIMARY OUTCOMES:
Cocaine abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Domenic Ciraulo, M.D., Principal Investigator — Boston University
Locations (6):
- United States (6):
  - Boston University Medical Center, Boston, Massachusetts
  - New York VA Medical Center, New York, New York
  - Cincinnati Addiction Research Center, Cincinnati, Ohio
  - Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania
  - RHD Professional Plaza 4, Dallas, Texas
  - UTHSCSA, San Antonio, Texas